CLINICAL TRIAL: NCT04565314
Title: ELICIT 2.0: Pilot Study of the Effect of Maternal Protein Supplementation During Lactation on Childhood Growth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Collaborators: Haydom Lutheran Hospital (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Mark D. DeBoer, MD, MSc., MCR, Professor of Pediatrics, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21967
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Growth Failure; Stunting; Malnutrition; Protein Malnutrition
Keywords: protein; breast feeding; eggs; Ready-to-eat food; infant; growth; Tanzania
MeSH Terms: conditions — Failure to Thrive; Growth Disorders; Malnutrition; Kwashiorkor; Breast Feeding

STUDY DESIGN:
Intervention Model Description: Participating mothers nursing children age 0-3 months at enrollment will receive 3 months of treatment with one packet of Plumpy'Mum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plumpy'Mum (Experimental): Mother/child dyads will be enrolled at child age 0-3 months and mothers will immediately begin consuming a packet of Plumpy'Mum (or similar protein food product) daily. Plumpy'Mum will be provided by the study team to the mother, who will consume this however she desires (i.e., alone or with other food). Intervention will continue for 3 months. The rational is that Plumpy'Mum consumption will improve the quality of the breast milk the child is consuming, contributing to improved growth over time. Growth will be compared to historical controls from prior studies in the area.
  Interventions: Dietary Supplement: Plumpy'Mum

INTERVENTIONS:
Dietary Supplement: Plumpy'Mum — Mothers will consume Plumpy'Mum (one packet daily) from enrollment (child age 0-3 months) for 3 months.

SUMMARY:
Haydom Global Health Research Center in north central Tanzania represents an important rural setting for performing high-quality medical research in sub-Saharan Africa. The region around Haydom is agricultural (predominantly maize-based), is resource-poor and has a high degree of stunting among local infants-with 70% stunting by 18 months in the MAL-ED study and 50% in the ELICIT study (for Early Life Interventions for Childhood Growth and Development In Tanzania). While the causes of this stunting are multifactorial, a potential contributor is early-life nutritional deficiencies, including inadequate dietary protein.

One likely source of low protein delivery to infants is from low intake among area mothers during lactation, with potential effects on breast milk protein content and child weight gain. The current study is a pilot study assessing our study team's ability to successfully deliver protein-containing food products (a balanced-energy protein supplement) to lactating mother is in the area and assessing whether consumption of these food products improves childhood growth in the 1st year of life. This is a pilot study because of the potential difficulties in distributing these products on a large scale for daily consumption. As such, we aim to demonstrate an effective distribution network, a means of assessing adherence, and measuring endpoints while gathering knowledge regarding community acceptance. The current pilot project will evaluate the effectiveness of distribution and adherence on approximately 100 mother/child dyads. If effective, a future project could involve a large enough sample to be powered to detect reasonable changes in linear growth. .

So, while the current proposal is not adequately powered to prove a hypothesis, the hypothesis underlying the study design is that daily protein supplementation delivered as a balanced protein product (Plumpy'mum) to lactating mothers for 3 months during the period from 0-6 months post-natal life will result in an increase in infant length-for-age Z-score (LAZ) by end of treatment. LAZ will be compared to controls from prior studies in the area.

DETAILED DESCRIPTION:
In severely under-resourced areas of the world, such as the Haydom area in Tanzania (TZ), poor nutrition continues contributes to worsened health-related outcomes including growth and cognitive development. Haydom Global Health Research Center at Haydom Lutheran Hospital in north central Tanzania represents an important rural setting for performing high-quality medical research in sub-Saharan Africa. Through ongoing work in the area around Haydom in the MAL-ED and ELICIT studies, we have been attempting to improve outcomes for children in an area of severe poverty, where there is considerable malnutrition and potential sequelae:

1. Growth deficits: Poor weight gain and linear growth failure in childhood are often seen as surrogates for overall health status; persistently poor growth has implications for future work potential and lower human capital. There was a high degree of stunting in the Haydom site of Tanzanian in the multi-country observational MAL-ED study, which found that the Haydom site had the highest prevalence of stunting among all the MAL-ED sites. This degree of stunting is likely multi-factorial, though one contributor is food availability, as rates of key factors such as birthweight vary significantly according to food availability. An interim analysis of data from our ongoing ELICIT study (for Early Life Interventions for Childhood

Developmental delays: Perhaps there is no more important outcome (with the exception of mortality) than the cognitive, social and emotional development of a population, with clear extensions to human capital, economic productivity and quality of life in communities. Indeed, many observational and interventional studies (including the current study) follow growth as an outcome because of its overall association with cognitive development. In MAL-ED assessments, TZ children had fewer words than seen among US children. The reasons for potential developmental delays are multifactorial, but again malnutrition may play an important role. Studies in other developing areas have demonstrated improved cognitive development following delivery of nutrition support.

Nutritional Causes of Poor Growth

While the causes of the stunting and developmental delays are multifactorial, a potential contributor is early-life nutritional deficiencies, including inadequate dietary protein. One likely source of low protein delivery to infants is from low intake among area mothers during lactation, with potential effects on breast milk protein content and child weight gain. Indeed, the first six months of life represents a critical phase of nutrition for the developing infant, in which all (or nearly all) nutrition is delivered through the mother's breast milk. However, it is not known whether protein supplementation during lactation in this setting would improve childhood growth and reduce stunting-or whether any improvements in growth would continue beyond the period of maternal supplementation.

Assessing the potential effect of mothers receiving protein supplementation-using a balanced energy protein supplement-on childhood growth and development would require an approach that incorporates an effective distribution network, a means of assessing adherence, and a thorough knowledge of community acceptance, as well as accurate measures of endpoints on a large enough sample to be powered to detect reasonable changes in linear growth. In order to assess the feasibility of this type of approach on a smaller scale (which could be later be expanded), the current pilot project will evaluate the effectiveness of distribution and adherence on approximately 100 mother/child dyads. If this experimental approach is feasible and shows promise, it is our hope to follow it with a larger study that offers more definitive evidence of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age >/= 18 years
* Current pregnancy or infant </= 3 months

Exclusion Criteria:

* Maternal inability to adhere to protocol
* Multiple gestation
* Significant birth defect
* Maternal allergy to peanut, milk or soy
* Lack of breast feeding at enrollment (and lack of intention to continue breast feeding at time of enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Family perception of Plumpy'Mum | at 3 months after enrollment
  Families will be queried about their impression of Plumpy'Mum

SECONDARY OUTCOMES:
Child weight-for-age Z-score (WAZ) after 3 months of Plumpy'Mum use | 3 months
  Child weight for WHO Z-score after 3 months of Plumpy'Mum use compared to historical controls
Child head circumference-for-age Z-score (HCZ) after 3 months of Plumpy'Mum use | 3 months
  Child head circumference for WHO Z-score after 3 months of Plumpy'Mum use compared to historical controls
Child mid-upper arm circumference-for-age Z-score (MUAC-Z) after 3 months of Plumpy'Mum use | 3 months
  Child mid-upper arm circumference Z-score after 3 months of Plumpy'Mum use compared to historical controls
Child length-for-age Z-score (LAZ) after 3 months of Plumpy'Mum use | 3 months
  Child length for WHO Z-score after 3 months of Plumpy'Mum use compared to historical controls
Adverse events | 3 months
  Number of adverse events in intervention arm, compared to historical controls
Maternal weight at 3 months | 3 months
  Maternal weight at 3 months compared to historical controls
Maternal mid-upper arm circumference-for-age Z-score (MUAC) at 3 months | 12 months
  Maternal mid-upper arm circumference at 3 months compared to historical controls

CONTACTS AND LOCATIONS:
Overall Officials: Mark D DeBoer, MD, MSc, MCR, Principal Investigator — University of Virginia
Locations (1):
- Haydom Lutheran Hospital, Mbulu, Manyara Region, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
We will assess platforms for sharing individual participant data following final data analysis.
Supporting Information: Study Protocol
Time Frame: Within 1 year after publication of results
Access Criteria: Contact PI to request